CLINICAL TRIAL: NCT05126615
Title: Contribution of Auriculotherapy in the Management of Mastectomy With Immediate Reconstruction by Latissimus Dorsi Flap (ATMAGD)
Acronym: ATMAGD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of recruitment
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018-A01108-47
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Mastectomy; Auriculotherapy
MeSH Terms: interventions — Auriculotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with auriculotherapy (Experimental): Mastectomy operated patient then, auriculotherapy
  Interventions: Drug: Auriculotherapy; Behavioral: Chronic Post-Surgical Pain evaluation
- Patient with placebo (Placebo Comparator): Mastectomy operated patient then, they received placebo
  Interventions: Behavioral: Chronic Post-Surgical Pain evaluation

INTERVENTIONS:
Drug: Auriculotherapy — Application of a bolus of 5 μ of liquid nitrogen via a cryospray on the auriculotherapy points A4, C18, D9, C9, DIX, H13, G14 and FXVII, chosen according to a neurophysiological reasoning taking into account the surgical intervention performed and innervation of the anatomical region affected by the intervention.
  Arms: Patients with auriculotherapy
Behavioral: Chronic Post-Surgical Pain evaluation — Different questionnaires :
  BPI : Brief Pain Inventory DN4

SUMMARY:
Over the past decade, more and more healthcare professionals are using auriculotherapy as a preventative and effective therapy for pain. This therapy is applied by odontologists, anesthetists, surgeons, etc., to alleviate chronic pain. The effects of auriculotherapy are known in particular in reducing preoperative anxiety, pain in cancer patients and postoperative pain.

The aim of this study is to assess the effectiveness of adding auriculotherapy to the standard global anesthetic protocol, compared to this single reference protocol, on the incidence at 3 months post-intervention of Chronic Post-Surgical Pain, in patients operated for a mastectomy with reconstruction immediate by latissimus dorsi flap.

ELIGIBILITY:
Inclusion Criteria:

* Women patient over 18 years-old
* Patient scheduled for a mastectomy with immediate reconstruction by latissimus dorsi flap with or without symmetrization on the contralateral breast.
* Patient affiliated or beneficiary of a social security scheme.
* Patient who has given her free and informed consent.
* Preoperative blood test showing no contraindication to the operation.

Exclusion Criteria:

* Refusal of the patient.
* No indication for auriculotherapy:
* Patient having a heavy treatment with neuroleptics,
* Or tricyclic antidepressants which interfere with the action of auriculotherapy.
* Patient undergoing long-term morphine treatment for chronic pain.
* Patient with unweaned opioid addiction.
* Chronic painful patient.
* Protected patient: Major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision; Hospitalized without consent.
* Pregnant, breastfeeding or parturient woman.
* Patient participating in another interventional study.
* Patient who had already participated in this study as part of first breast surgery.
* Patient receiving regular care by auriculotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Presence, or not, of Chronic Post-Surgical Pain (DCPC) | 3 months
  DCPC noted during the clinical examination of the 3rd postoperative month :
  - score obtained at BPI : Brief Pain Inventory (9 items : many items with answers between 0 and 10)
Presence, or not, of Chronic Post-Surgical Pain (DCPC) | 3 months
  DCPC noted during the clinical examination of the 3rd postoperative month :
  - score obtained at DN4 (neuropathic pain) : 4 different items

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Paul d'Egine, Champigny-sur-Marne, France